CLINICAL TRIAL: NCT04563169
Title: Video Consultation as an Adequate Alternative to Face-to-face Consultations in CPAP Use for Patients With Obstructive Sleep Apnea: Randomized Controlled Trial.
Brief Title: Video Consultation in CPAP for Patients With Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2018-1165
Record Dates: First submitted 2020-09-16; First posted 2020-09-24 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Obstructive Sleep Apnea
Keywords: Video consultation; E-Health; CPAP; Randomized Controlled Trial
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video consultation (Experimental): Patients in the video consultation group will receive video consultations.
  Interventions: Other: Video consultation
- Face-to-Face consultation (No Intervention): Patients in the usual care group will receive face-to-face consultations.

INTERVENTIONS:
Other: Video consultation — The first video consultation with a nurse was planned one week after start with CPAP. Three focus points were discussed during the consultations: 1) adherence (>6 hours per night); 2) rest AHI < 5 (or <10 if age >70), and 3) (improvements in) complaints. If these objectives were achieved after one week, a new consultation was planned three weeks later (four weeks after start). As long as these objectives were not achieved, video consultations were planned weekly (until after four weeks).
  Arms: Video consultation

SUMMARY:
The objective of this study is to evaluate the effects of video consultation versus face-to-face consultation for patients with obstructive sleep apnea on patients' CPAP use (minutes/per night), self-efficacy, risk outcomes, outcome expectancies, experiences with technology and, patients' and nurses' satisfaction.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the effects of video consultation versus face-to-face consultation for patients with obstructive sleep apnea on patients' CPAP use (minutes/per night), self-efficacy, risk outcomes, outcome expectancies, experiences with technology and, patients' and nurses' satisfaction.

This study is a non-blinded randomized controlled trial with an intervention group (video consultations) and a usual care group (face-to-face consultations), with assessements after 1, 2, 3, 4, 12 and 24 weeks.

Patients were recruited from a large teaching hospital (Rijnstate, hospital), and included from January 2, 2019 until June 26, 2019.In total, 140 patients were randomized, (1:1 allocation).

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* Diagnosed with obstructive sleep apnea
* AHI > 15
* Requiring CPAP treatment
* No history of CPAP treatment
* Having access to a tablet or smartphone
* Proficiency of the Dutch language

Exclusion Criteria:

* Psychiatric or cognitive disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2019-12-09 (Actual); Study Completion 2019-12-09 (Actual)

PRIMARY OUTCOMES:
CPAP use | Week 1 through week 4
  Continuous Airway Pressure use (minutes/night), extracted from Encore Anywhere.
CPAP use | Week 4 through week 12
  Continuous Airway Pressure use (minutes/night), extracted from Encore Anywhere.

SECONDARY OUTCOMES:
CPAP adherence | Week 1 through week 4
  CPAP use for at least 5 nights per week for at least 4 hours per night. Extracted from Encore Anywhere.
CPAP adherence | Week 4 through week 24
  CPAP use for at least 5 nights per week for at least 4 hours per night. Extracted from Encore Anywhere.
Self-efficacy | Baseline
  Self-Efficacy Measure for Sleep Apnea questionnaire. Items were rated with a 4 point scale, varying from 1 (not at all true) to 4 (very true).
Self-efficacy | Week 4
  Self-Efficacy Measure for Sleep Apnea questionnaire. Items were rated on a 4 point scale, varying from 1 (not at all true) to 4 (very true).
Outcome expectancies | Baseline
  Assessed with Self-Efficacy Measure for Sleep Apnea questionnaire. Items were rated on a 4 point scale, varying from 1 (not at all true) to 4 (very true).
Outcome expectancies | Week 4
  Self-Efficacy Measure for Sleep Apnea questionnaire. Items were rated on a 4 point scale, varying from 1 (not at all true) to 4 (very true).
Risk perception | Baseline
  Self-Efficacy Measure for Sleep Apnea questionnaire. Items were rated on a 4 point scale, varying from 1 (very low) to 4 (very high).
Risk perception | Week 4
  Assessed with Self-Efficacy Measure for Sleep Apnea questionnaire. Items were rated on a 4 point scale, varying from 1 (very low) to 4 (very high).
Expectations with video consultation | Baseline
  Questions based on constructs of the Unified Theory of Acceptance and Use of Technology. Items were rated on a 7 point scale, varying from 1 (totally disagree) to 7 (totally agree).
Experiences video consultation | Week 4
  Questions based on constructs of the Unified Theory of Acceptance and Use of Technology (intervention group only). Items were rated on a 7 point scale, varying from 1 (totally disagree) to 7 (totally agree).
Satisfaction patients | Week 4
  Questionnaires were used to assess satisfaction about consultations, number of consultations, received information, satisfaction with video consultation (intervention group only) and suggestions for improvement of the use of video consultation (open ended question). Items were rated on a 5 point scale, varying from 1 (totally disagree) to 5 (totally agree). Overall satisfaction was rated on a scale varying from 1 (not satisfied) to 10 (very satisfied).
Satisfaction patients | After intervention completion, up to 8 months (after start).
  Satisfaction with video consultation, benefits (eg, time and efficiency) and integration in work process. Items were rated on a 5 point scale, varying from 1 (totally disagree) to 5 (totally agree). Overall satisfaction was rated on a scale varying from 1 (not satisfied) to 10 (very satisfied). Suggestions for improvement were assessed using an open question

OTHER OUTCOMES:
Sex | Baseline
  Female/male
Age | Baseline
  Age (years)
Education | Baseline
  Education
Living together with a partner | Baseline
  Living together wit a partner (yes/no).
Internet use | Baseline
  Internet use (duration) varying from less than six months until more than 3 years.

CONTACTS AND LOCATIONS:
Overall Officials: Wim van Harten, Principal Investigator — Rijnstate Hospital
Locations (1):
- Rijnstate, Arnhem, Netherlands

REFERENCES:
- [Derived] Kooij L, Vos PJ, Dijkstra A, Roovers EA, van Harten WH. Video Consultation as an Adequate Alternative to Face-to-Face Consultation in Continuous Positive Airway Pressure Use for Newly Diagnosed Patients With Obstructive Sleep Apnea: Randomized Controlled Trial. JMIR Form Res. 2021 May 11;5(5):e20779. doi: 10.2196/20779. PMID 33973866

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-12): https://cdn.clinicaltrials.gov/large-docs/69/NCT04563169/Prot_SAP_000.pdf